CLINICAL TRIAL: NCT01415960
Title: Efficacy and Safety of a New Leuprolide Acetate 22.5 mg Depot Formulation in the Treatment of Prostate Cancer
Brief Title: Efficacy and Safety of Leuprolide Acetate 22.5 mg Depot in Treatment of Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GP-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GP/C/05/PRO
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2016-11

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; androgen deprivation therapy.; Leuprolide Acetate Depot Formulation; Pharmacokinetics; testosterone; serum luteinizing hormone; follicle-stimulating hormone; prostate-specific antigen
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Leuprolide acetate 22.5 mg depot (Experimental): Leuprolide acetate 22.5 mg depot administered twice, 3 months apart
  Interventions: Drug: Leuprolide acetate 22.5 mg depot, GP-Pharm SA

INTERVENTIONS:
Drug: Leuprolide acetate 22.5 mg depot, GP-Pharm SA — Administered by im injection, twice during the study, three months apart

SUMMARY:
Some patients with prostate cancer benefit from androgen deprivation therapy which reduces levels of testosterone. Leuprolide is a synthetic Luteinizing hormone releasing hormone (LHRH) analogue which upon administration can decrease testosterone levels to ≤0.5 ng/mL. Leuprolide Acetate 22.5 mg Depot is a microencapsulated formulation of leuprolide which is released slowly over time and effectively reduces testosterone levels in many patients to ≤0.5 ng/mL for up to three months. In this study Leuprolide acetate 22.5 mg Depot will be administered by intramuscular injection twice over a period of 6 months. The proportion of patients with testosterone ≤0.5 ng/mL evaluated over a period of 168 days.

DETAILED DESCRIPTION:
This in an open-label, multicenter, multiple-dose investigation of 2 doses of leuprolide acetate 22.5 mg administered with a 3-month interval to patients with histologically proven carcinoma of prostate who might benefit from medical androgen deprivation therapy. A total of up to 160 male patients will receive their first single intramuscular injection of leuprolide acetate 22.5 mg on Day 0 (after baseline assessment) and then after 3 months (Day 84). The study duration will be 6 months. Thirty(30) patients will be screened per protocol and enrolled at selected centers to form the PK cohort. The PK/PD analysis will be performed using plasma specimens from the first 20 of 30 patients enrolled in the study (and included in the PK/PD cohort). Patients not belonging to the PK cohort will be screened and enrolled per protocol and will follow the same study schedule as those enrolled in the PK portion of the study, except they will provide only sparse PK sampling.

ELIGIBILITY:
Main selection criteria:

Patients with histologically documented prostate cancer who might benefit from medical androgen deprivation therapy (i.e., reduction of androgen levels) will be considered for enrollment in the study if they meet the following criteria:

Inclusion Criteria:

1. Males ≥18 years of age
2. Patients with histologically documented prostate carcinoma who might benefit from medical androgen deprivation therapy.
3. Life expectancy of at least 1 year.
4. WHO/ECOG performance status of 0, 1, or 2.
5. Adequate renal function at Screening as defined by serum creatinine ≤1.6 times the upper limit of normal (ULN) for the clinical laboratory.
6. Adequate and stable hepatic function as defined by bilirubin ≤1.5 times the ULN and transaminases (i.e., aspartate aminotransferase, alanine aminotransferase) ≤2.5 times the ULN for the clinical laboratory at Screening.
7. Ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to cooperate with the investigator and to comply with the requirements of the entire study.
8. Following receipt of verbal and written information about the study,the patient must provide signed informed consent before any study related activity is carried out.

Exclusion Criteria:

1. Evidence of brain metastases, in the opinion of the investigator, taking into account medical history, clinical observations, and symptoms (rationale: to minimize possibility of serious acute flare reactions that would necessitate concomitant administration of other drugs).
2. Evidence of spinal cord compression, in the opinion of the investigator, taking into account medical history, clinical observations, and symptoms (rationale: see rationale in criterion 1).
3. Evidence of severe urinary tract obstruction with threatening urinary retention, in the opinion of the investigator, taking into account medical history, clinical observations, and symptoms (rationale: see rationale in criterion 1).
4. Presence of any tumor in the immediate vicinity that could cause spinal cord compression, in the opinion of the investigator, taking into account medical history and clinical observations (rationale: see rationale in criterion 1).
5. Excruciating, severe pain from extensive osseous deposits, taking into account medical history, clinical observations, and symptoms (rationale: see rationale in criterion 1).
6. Testosterone levels <1.5 ng/mL at Screening, This testosterone level will be locally determined at the laboratory of each clinical site (rationale: to ensure that all patients have normal baseline testosterone levels).
7. Previous androgen ablative therapy lasting more than 6 months, such as LHRH analogues (e.g., Leuprolide acetate, Goserelin, Buserelin) or antagonists (degarelix). Also, therapy must have not occurred within 12 months before the screening visit. Any prior ADT must have not exceeded 6 months of therapy.
8. Previous treatment with androgen-receptor blockers, such as Bicalutamide, Flutamide, Megestrol acetate, Ciproterone will only be allowed after a 3 month washout prior to the screening visit (rationale: these therapies alter a patient's androgenic hormonal response for a sustained period).
9. Previous orchiectomy, adrenalectomy, or hypophysectomy (no washout allowed) (rationale: these therapies could have altered a patient's androgenic hormonal response).
10. Previous prostatic surgery (e.g., radical prostatectomy, transurethral resection of the prostate) within 2 weeks before Baseline (rationale: these therapies could have altered a patient's androgenic hormonal response and/or adverse reaction profile).
11. Previous local therapy to the primary tumor with a curative attempt other than surgery (external beam radiotherapy, brachytherapy, thermotherapy, cryotherapy) within 2 weeks before Baseline (rationale: these therapies could have altered a patient's adverse reaction profile).
12. Previous cancer systemic therapy such as chemotherapy, immunotherapy (e.g., antibody therapies, tumor vaccines), biological response modifiers (e.g., cytokines).
13. Any investigational drug within 5 half-lives of its physiological action or 3 months, whichever is longer, before Baseline (rationale: to prevent adverse effects of another drug being attributed to study drug and to prevent potential interactions).
14. Administration of 5-α-reductase inhibitors (Finasteride, Dutasteride) within 3 months before Baseline (rationale: alters PSA levels and androgen metabolism of the prostate cells). Prior use of 5-α-reductase inhibitors will be allowed with a 3 month washout.
15. Over-the-counter or alternative medical therapies that have an estrogenic or antiandrogenic effect (i.e., PC-SPES, saw palmetto, Glycyrrhiza, Urinozinc, dehydroepiandrosterone) within the 3 months before Baseline.
16. Hematological parameters (red blood cells, total and differential white blood cell count, platelet count, hemoglobin, hematocrit) outside 20% of the ULN or lower limits of normal for the clinical laboratory at Screening (rationale: to render potential study drug-related laboratory abnormalities easier to observe).
17. Coexistent malignancy, in the opinion of the investigator (rationale: to decrease possibility of disease-caused or associated therapy-caused adverse effects being attributed to study drug).
18. Uncontrolled congestive heart failure, myocardial infarction or a coronary vascular procedure (e.g., balloon angioplasty, coronary artery bypass graft) or significant symptomatic cardiovascular disease(s) within 6 months before Baseline; resting uncontrolled hypertension (≥160/100 mm Hg) or symptomatic hypotension within 3 months before Baseline (rationale: to decrease possibility of disease-caused or associated therapy-caused adverse effects being attributed to study drug).
19. Venous thrombosis within 6 months of Baseline (rationale: influencing testosterone levels may be associated with increased likelihood of deep venous thrombosis).
20. Uncontrolled diabetes, in the opinion of the investigator (rationale:

    patients with uncontrolled diabetes need to compensate the metabolic disorder before treatment with LHRH analogues).
21. History of drug and/or alcohol abuse within 6 months of Baseline (rationale: these patients are likely to have numerous medical abnormalities and are unlikely to comply with protocol).
22. Serious concomitant illness(es) or disease(s) (e.g., hematological, renal, hepatic, respiratory, endocrine, psychiatric) that may interfere with, or put patients at additional risk for, their ability to receive the treatment outlined in the protocol (rationale: to decrease possibility of disease-caused or associated therapy-caused adverse effects being attributed to study drug).
23. Patients on anticoagulative therapy including warfarin (Coumadin®), Dabigatran Etexilate (Pradaxa®) and heparin. Those patients on low-dose, low-molecular weight heparin may be enrolled in the study (rationale: to decrease possibility of disease-caused or associated therapy-caused adverse effects being attributed to study drug). Plavix and Aspirin are allowed for cardiac prophylaxis as long as all inclusion/exclusion criteria are met concerning coagulation parameters and thromboembolic history. Special care to avoid hematoma at the injection site must be observed.
24. Abnormal coagulation studies (prothrombin time [PT]/partial thromboplastin time [PTT]) at Baseline.
25. History of serious bleeding on injections, an elevated INR, concomitant medications or any other condition (i.e. significant thrombocytopenia) that in opinion of the investigator would render the subject at risk of significant bleeding with injections.
26. Blood donations/losses within 2 months of Baseline, apart from previous prostatic surgery patients (see exclusion 10 [rationale: to avoid excessive blood donations]).
27. Known hypersensitivity to GnRH, GnRH agonists, including any LHRH analogues, or any excipients of the study formulation (rationale: to minimize hypersensitivity reaction to study drug).
28. History of Immunization (within 4 weeks of Baseline) and specifically flu shots (within 1 week of Baseline or 1 week before and after study drug administration) (Rationale: to decrease the possibility of non treatment-related AEs being attributed to study drug).
29. Skin disease that would interfere with injection site evaluation.
30. Men not willing to use appropriate birth control methods such as surgical sterilization or barrier contraception or men with partners of child bearing potential not willing to use appropriate birth control methods, such as surgical sterilization, hormonal birth control (partner), an intrauterine device (partner) or double-barrier method for the entire study period.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Genesis Research, San Diego, California
  - Atlantic Urological Associates, Daytona Beach, Florida
  - Urology Health Team, Ocala, Florida
  - Winter Park Urology Associates, PA, Orlando, Florida
  - Coastal Medical Center, Sarasota, Florida
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Idaho Urologic Institute, Meridian, Idaho
  - First Urology, Jeffersonville, Indiana
  - Mid Atlantic Clinical Research, Greenbelt, Maryland
  - Premier Urology Associates, LLC, Lawrenceville, New Jersey
  - The Urological Institute of Northeastern New York, Albany, New York
  - Brooklyn Urology Research Group, Brooklyn, New York
  - Manhattan Medical Research, New York, New York
  - The Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - Staten Island Urological Research, PC, Staten Island, New York
  - PMG Research of Wilmington, Wilmington, North Carolina
  - PMG Research of Winston Salem, Winston-Salem, North Carolina
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Urology Health Specialists, LLC, Bryn Mawr, Pennsylvania
  - Greenville Health System, Greer, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, PC, Nashville, Tennessee
  - Urology San Antonio Research, PA, San Antonio, Texas
  - Urology of Virginia, Virginia Beach, Virginia
  - Seattle Urology Research Center, Burien, Washington

REFERENCES:
- [Derived] Shore ND, Guerrero S, Sanahuja RM, Gambus G, Parente A. A New Sustained-release, 3-Month Leuprolide Acetate Formulation Achieves and Maintains Castrate Concentrations of Testosterone in Patients With Prostate Cancer. Clin Ther. 2019 Mar;41(3):412-425. doi: 10.1016/j.clinthera.2019.01.004. Epub 2019 Feb 8. PMID 30929678

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Leuprolide Acetate 22.5 mg Depot
Started | 163
ITT | 161
PK Subgroup | 30
Completed | 151 (Patients completed Study (151) Per protocol Patients (146))
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | Leuprolide Acetate 22.5 mg Depot
Number analyzed (Participants) | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 161
Region of Enrollment [Number; unit: participants]
  United States | 161

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Chemical Castration (Defined as Testosterone Levels ≤ 0.5 ng/mL) at Days 28, 84, and 168.
Description: The primary endpoint was testosterone ≤ 0.5 ng/mL assessed on Days 28, 84, and 168. Thereby, maintenance of castration was to be demonstrated through Day 168 with no missing data at these key time points, unless the missing data were due to an event unrelated to the study drug (ITT patients).
Time Frame: 168 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Leuprolide Acetate 22.5 mg Depot: Leuprolide acetate 22.5 mg depot administered twice, 3 months apart.
  Leuprolide acetate 22.5 mg depot, GP-Pharm SA: Administered by im (intramuscular) injection, twice during the study, three months apart.
Arm/Group | Leuprolide Acetate 22.5 mg Depot
Number analyzed (Participants) | 161
percentage of participants | 98.1 [94.7 to 99.6]

2. Secondary Outcome: Determination of Serum Luteinizing Hormone (LH)
Description: For purposes of calculating summary statistics, any concentration values Below Limit of Quantification (BLQ) were to be assigned ½ the Low Limit of Quantification (LLOQ) (LLOQ=2.00). If the calculated mean, median or minimum value at a time point was less than LLOQ, "BLQ" is presented. In addition, since a high proportion of BLQ values may affect the Standard Deviation (SD); if more than 50% of values were imputed, then no mean or median was calculated for that time point.
Time Frame: 168 days
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Leuprolide Acetate 22.5 mg Depot
Number analyzed (Participants) | 161
mIU/mL
  Baseline | 7.24 (6.48)
  Day 28 | 1 (2.79)
  Day 168 | 1 (0.92)

3. Secondary Outcome: Follicle-stimulating Hormone (FSH)
Description: For purposes of calculating summary statistics, any concentration values Below Limit of Quantification (BLQ) were to be assigned ½ the Low Limit of Quantification (LLOQ) (LLOQ=3.66). If the calculated mean, median or minimum value at a time point was less than LLOQ, "BLQ" is presented. In addition, since a high proportion of BLQ values may affect the Standard Deviation (SD); if more than 50% of values were imputed, then no mean or median was to be calculated for that time point.
Time Frame: 168 days
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Leuprolide Acetate 22.5 mg Depot
Number analyzed (Participants) | 161
mIU/mL
  Baseline | 15.14 (13.46)
  Day 28 | 1 (1.44)
  Day 168 | 5.80 (3.62)

4. Secondary Outcome: Prostate-specific Antigen (PSA) Concentrations
Description: For purposes of calculating summary statistics, any concentration values Below Limit Quantification (BLQ) were to be assigned ½ the Low Limit Quantification (LLOQ) (LLOQ=0.36). If the calculated mean, median or minimum value at a time point was less than LLOQ, "BLQ" is presented. In addition, since a high proportion of BLQ values may affect the Standard Deviation (SD); if more than 50% of values were imputed, then no mean or median was calculated for that time point.
Time Frame: 168 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Leuprolide Acetate 22.5 mg Depot
Number analyzed (Participants) | 161
ng/mL
  Baseline | 44.36 (165.81)
  Day 168 | 2.37 (10.30)

5. Secondary Outcome: Determination of Leuprolide Cmax
Description: Leuprolide Pharmacokinetic Parameters (PK Population).
Time Frame: Cmax1: 0, 1 and 4 hours post-dose on Day 0 and once on Days 2, 14, 28, 56; Cmax2: 0, 1 and 4 hours post-dose on Day 84 and once on Days 86, 112 and 168.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Leuprolide Acetate 22.5 mg Depot
Number analyzed (Participants) | 30
ng/mL
  Day 0/Dose 1 Cmax | 46.79 (18.008)
  Day 84/Dose 2 Cmax | 48.30 (18.557)

6. Secondary Outcome: Safety Endpoints
Description: The WHO/ECOG, bone pain, urinary pain and urinary symptoms data reported are the most frequent percentage at the assessment time.
  * The WHO/ECOG performance status was summarized using the 0 to 4 WHO/ECOG performance status scale. (0= fully active, able to carry on all pre-disease performances without restriction).
  * Bone pain, urinary pain and urinary symptoms were determined using a 10-point scale (1= no pain/symptoms, 10= worst pain/symptom imaginable).
Time Frame: 168 Days
Population: Safety endpoints adverse events (AEs), local tolerability, vital signs, performance status, bone pain, urinary pain, and urinary symptoms, occurrence of hot flushes and clinical laboratory and electrocardiogram (ECG) results.
Measure: Number; unit: percentage of participants
Arm/Group | Leuprolide Acetate 22.5 mg Depot
Number analyzed (Participants) | 161
percentage of participants
  Baseline WHO/ECOG Score 0 (n=161) | 83.9
  Day 168 WHO/ECOG Scores 0 (n=152) | 82.9
  Baseline Bone Pain score 1 (n=161) | 95.0
  Day 168 Bone Pain score 1 (n=152) | 94.1
  Baseline Urinary Pain score 1 (n=161) | 98.8
  Day 168 Urinary Pain Score 1 (n=152) | 97.4
  Baseline Urinary Symptoms score 1 (n=161) | 87.6
  Day 168 Urinary Symptoms score 1 (n=152) | 89.5

7. Secondary Outcome: Determination of Leuprolide Tmax
Description: Leuprolide Pharmacokinetic Parameters (PK Population).
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Leuprolide Acetate 22.5 mg Depot
Number analyzed (Participants) | 30
day
  Day 0/Dose 1 Tmax | 0.07 (0.051)
  Day 84/Dose 2 Tmax | 0.08 (0.056)

ADVERSE EVENTS:
Arm/Group | Leuprolide Acetate 22.5 mg Depot
Serious Adverse Events (participants affected / at risk) | 12/163
Other Adverse Events (participants affected / at risk) | 141/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprolide Acetate 22.5 mg Depot (N=163)
CONGESTIVE HEART FAILURE (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
DIARRHEA (Gastrointestinal disorders) | 1
INCARCERATED INGUINAL HERNIA (Gastrointestinal disorders) | 1
RECTAL BLEEDING (Gastrointestinal disorders) | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1
PNEUMONIA (Infections and infestations) | 1
FALL (Injury, poisoning and procedural complications) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1
BENIGN NEOPLASM OF BLADDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SYNCOPE (Nervous system disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leuprolide Acetate 22.5 mg Depot (N=163)
TEAE Related Injection site pain (General disorders) | 15 (16)
TEAE Related Fatigue (General disorders) | 16 (19)
TEAE Related Hot Flushes (Vascular disorders) | 126 (146)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information from the trial is property of the Sponsor and the PI has no right on it except the prior writing authorization of the sponsor